CLINICAL TRIAL: NCT02106767
Title: The Effects of Single-Dose Rifampin on the Pharmacokinetics of Rosuvastatin in Healthy White and Asian Volunteers
Brief Title: The Effects of Rifampin on the Pharmacokinetics of Rosuvastatin
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 14-12970
Record Dates: First submitted 2014-04-03; First posted 2014-04-08 (Estimated); Last update posted 2020-01-23 (Actual); Status verified 2020-01

CONDITIONS: Healthy
Keywords: rosuvastatin; rifampin; pharmacokinetics; drug interaction; healthy volunteer; drug transporter; Asian; White
MeSH Terms: interventions — Rosuvastatin Calcium; Rifampin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Rosuvastatin (Active Comparator)
  Interventions: Drug: Rosuvastatin
- Rifampin plus rosuvastatin (Experimental)
  Interventions: Drug: Rosuvastatin plus rifampin

INTERVENTIONS:
Drug: Rosuvastatin — Rosuvastatin 20mg po x1
  Other Names: Crestor
  Arms: Rosuvastatin
Drug: Rosuvastatin plus rifampin — Rifampin 600mg IV infused over 30 minutes followed by rosuvastatin 20mg PO x1
  Other Names: Crestor; Rifadin; Rifampicin
  Arms: Rifampin plus rosuvastatin

SUMMARY:
The effect of transporter inhibition by rifampin on the pharmacokinetics of rosuvastatin will be studied in clinical trial in White and Asian healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Asian volunteers of Han-Chinese/Japanese/Korean descent whose parents and grandparents are Han-Chinese/ Japanese/ Korean.
* Healthy Caucasian volunteers of White/Caucasian/European-born descent whose parents and grandparents are White/Caucasian/European.
* Male or female, ages 18-65 years old, with no current medical conditions or active diagnoses as determined by the study doctor based on history, physical exam, and laboratory evaluations.
* Subjects who take no other medications two weeks prior to the study and during the time course of the study including prescription medications, over-the-counter medications, dietary supplements, or drugs of abuse.
* Subjects with the following genotype: SLCO1B1*1a and ABCG2 421CC.
* Subjects able to maintain adequate birth control during the study independent of hormonal contraceptive use.
* Subjects able to abstain from grapefruit, grapefruit juice, oranges, orange juice, caffeinated beverages and/or alcoholic beverages from 7am the day before the study to completion of that study day.
* Participants determined to have normal liver and kidney function as measured at baseline
* BMI between 18.0 - 30 kg/m2
* Subjects capable of fasting from food and beverages at least 8 hours prior to medication dosing.
* Be able to read, speak, and understand English.
* Subjects capable of providing informed consent and completing the requirements of the study.

Exclusion Criteria:

* Subjects with active medical problems
* Subjects on chronic prescription or OTC medication that cannot be stopped 2 weeks prior to and during the study.
* Subjects incapable of multiple blood draws (HCT < 30mg/dL)
* Subjects with a history of rhabdomyolysis
* Subjects with a history of drug-related myalgias
* Subjects with a history or diagnosis of hemorrhagic tendencies or blood dyscrasias
* Subjects with a history of GI bleed or peptic ulcer disease
* Subjects who smoke tobacco or have ongoing alcohol or illegal drug use
* Subjects who are pregnant, lactating, or trying to conceive during the study period
* Subjects allergic to rosuvastatin or rifampin or any known component of the medications
* Anyone who in the opinion of the study investigators is unable to do the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2014-11; Primary Completion 2016-08-07 (Actual); Study Completion 2016-08-07 (Actual)

PRIMARY OUTCOMES:
Area-under-the-concentration curve (AUC) of rosuvastatin | Blood samples collected over a 48 hour period

SECONDARY OUTCOMES:
Maximum plasma concentration (Cmax) of rosuvastatin | 0, 0.5, 1, 1.5, 2, 3, 4, 6, 9, 12, 24, 32, and 48 hours post-dose
Time to concentration maximum (Tmax) of rosuvastatin | 0, 0.5, 1, 1.5, 2, 3, 4, 6, 9, 12, 24, 32, and 48 hours post-dose

CONTACTS AND LOCATIONS:
Overall Officials: Leslie Z Benet, PhD, Principal Investigator — University of California, San Francisco; Lynda Frassetto, M.D., Principal Investigator — University of California, San Francisco
Locations (1):
- CTSI Clinical Research Center, UCSF, San Francisco, California, United States